CLINICAL TRIAL: NCT00343005
Title: Double-Blind, Randomized, Controlled, Phase 1 Study of the Safety and Immunogenicity of AMA1-C1/Alhydrogel Vaccine for Plasmodium Falciparum Malaria, in Semi-Immune Adults in Doneguebougou, Mali
Brief Title: Experimental Vaccine for Malaria in Adults in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999904175; 04-I-N175
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-01-22

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Blood-Stage; Investigational; Endemic; Malaria; Vaccine
MeSH Terms: conditions — Malaria, Falciparum; Burkitt Lymphoma; Malaria

INTERVENTIONS:
Biological: AMA1-C1
Drug: AMA1-C1/alhydrogel Malaria Vaccine

SUMMARY:
This study will determine the highest dose of an experimental vaccine called AMA1-C1 that can safely be given to adults exposed to malaria. Malaria affects about 300 million to 500 million people worldwide each year, causing from 2 million to 3 million deaths, mostly among children under 5 years of age in sub-Saharan Africa. It is the leading cause of death and illness among the general population of Mali in West Africa. Increasing drug resistance to the malaria parasite, as well as widespread resistance of mosquitoes (the insects that transmit the parasite) to pesticides are reducing the ability to control malaria through these strategies. A vaccine that could reduce illness and death from malaria would be a valuable new resource in the fight against this disease. AMA1-C1 is an experimental vaccine developed by the NIAID. Early tests of AMA1-C1 in 30 healthy people in the United States found no serious harmful side effects of the vaccine. This study will look at the effect of AMA1-C1 in people in Mali who have been exposed to malaria.

Residents of Don gu bougou, Mali, who are between 18 and 45 years of age and are in general good health may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, and urine pregnancy test for women.

Participants are randomly assigned to receive three injections (shots) of either the experimental malaria vaccine or a hepatitis B vaccine that is approved and used in Mali. All shots are given in an upper arm muscle. After the first shot, the second is given 1 month later, and the third is given 12 months after the first. Subjects receiving AMA1-C1 will get one of three different doses - low, medium, or high - to find the dose that is safest and gives the best antibody response to the vaccine. After each shot, participants remain in the clinic for 30 minutes for observation. They return to the clinic 1, 2, 3, 7, and 14 days after each shot for a physical examination and to check for side effects. Blood samples are drawn before each shot and at selected return clinic visits to check for side effects and to measure the effect of the vaccine.

During the rainy seasons after the second and third vaccinations, subjects come to the clinic once a month for an examination and a blood test. During the dry season, subjects come to the clinic 3 months before the last shot is given for an examination and blood test. Additional blood tests may be done on participants who develop malaria.

If found to be safe in adults, further studies with this vaccine will be done in children exposed to malaria, as it is children who bear the brunt of this disease.

DETAILED DESCRIPTION:
The purpose of this Phase 1 clinical trial is to evaluate the safety and immunogenicity of the Plasmodium falciparum malaria vaccine AMA1-C1/Alhydrogel, in healthy malaria-exposed adult volunteers. Between 2-3 million deaths occur each year as a result of malaria. Most of these deaths are a result of P. falciparum malaria, in children under five years of age, in sub-Saharan Africa. A safe and effective vaccine that would reduce both morbidity and mortality secondary to P. falciparum would be a valuable resource in the fight against this disease. The apical membrane antigen 1 (AMA1) is a surface protein expressed during the asexual blood stage of P. falciparum that is thought to play a role in parasite invasion of erythrocytes. Clinical symptoms of malaria in humans are due to the asexual blood stage. Therefore, this vaccine was designed to protect an individual from illness due to the asexual stage of P. falciparum infection by inhibiting parasite invasion of erythrocytes. The AMA1-C1/Alhydrogel vaccine preparations to be studied contain an equal mixture of AMA1 from two different clones of Plasmodium falciparum (FVO and 3D7), both produced separately as recombinant proteins expressed by Pichia pastoris (AMA1 FVO and AMA1 3D7). This vaccine has been tested in one clinical trial of 30 malaria-unexposed human adults in the United States and no clinically significant risks have been identified. The study will be conducted in Don gu bougou, Mali, and will be a blinded, randomized and controlled trial that will evaluate three dose levels of AMA1-C1 (5 micro g, 20 micro g, 80 micro g). Fifty-four healthy male and non-pregnant female volunteers ages 18 to 45 will be enrolled. Eighteen volunteers will be assigned to each of the three dose groups. Within each group, twelve volunteers will be randomized to receive either a 5 micro g, 20 micro g, or 80 micro g dose of AMA1-Cl/Alhydrogel and 6 will be randomized to receive the tetanus toxoid vaccine. Immunizations will be administered by intramuscular injection on months 0, 1, and 12. The groups will be staggered such that adequate safety evaluation can be performed prior to dose escalation. The duration of the study is 18 months per volunteer. The primary objective of this trial is to determine the frequency and severity of vaccine-related adverse events for each dose. The secondary objective is to determine the dose that generates the highest serum antibody levels to AMA1 antigen at Day 42.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males or females between 18 and 45 years, inclusive.

Known residents of the village of Doneguebougou, Mali.

Good general health as determined by means of the screening procedure.

Available for the duration of the trial (78 weeks).

Willingness to participate in the study as evidenced by signing the informed consent document.

EXCLUSION CRITERIA:

Pregnancy as determined by a positive urine beta-hCG (if female).

Participant and her spouse are unwilling to use reliable contraception methods up until one month following the third immunization (if female).

Currently lactating and breast-feeding (if female).

Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, chronic infectious or renal disease by history, physical examination, and/or laboratory studies including urinalysis.

Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.

Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25 times the upper limit of normal of the testing laboratory).

Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing).

Laboratory evidence of hematologic disease (absolute leukocyte count less than 3000/mm(3) or greater than 13.5 x 10(3)/mm(3); hemoglobin less than 0.9 times the lower limit of normal of the testing laboratory, by sex; absolute lymphocyte count less than 1000/mm(3); or platelet count less than 120,000/mm(3)).

Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.

Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.

History of a severe allergic reaction or anaphylaxis.

Severe asthma (emergency room visit or hospitalization within the last 6 months).

Positive ELISA for HCV.

Positive HBsAg by ELISA.

Known immunodeficiency syndrome.

Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study or while the study is ongoing.

Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.

History of a surgical splenectomy.

Receipt of blood products within the past 6 months.

Previous receipt of an investigational malaria vaccine.

History of a known allergy to nickel.

Previous receipt of a primary series of any Hepatitis B vaccine.

History of known allergy to yeast.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54
Dates: Start 2004-04-23; Study Completion 2008-01-22

CONTACTS AND LOCATIONS:
Locations (1):
- Malaria Research and Training Center (MRTC), Bamako, Mali

REFERENCES:
- [Background] Crewther PE, Culvenor JG, Silva A, Cooper JA, Anders RF. Plasmodium falciparum: two antigens of similar size are located in different compartments of the rhoptry. Exp Parasitol. 1990 Feb;70(2):193-206. doi: 10.1016/0014-4894(90)90100-q. PMID 2404781
- [Derived] Dicko A, Diemert DJ, Sagara I, Sogoba M, Niambele MB, Assadou MH, Guindo O, Kamate B, Baby M, Sissoko M, Malkin EM, Fay MP, Thera MA, Miura K, Dolo A, Diallo DA, Mullen GE, Long CA, Saul A, Doumbo O, Miller LH. Impact of a Plasmodium falciparum AMA1 vaccine on antibody responses in adult Malians. PLoS One. 2007 Oct 17;2(10):e1045. doi: 10.1371/journal.pone.0001045. PMID 17940609